CLINICAL TRIAL: NCT04601259
Title: A Prospective, Randomized, Controlled, Open-labelled Investigation to Assess Performance and Safety of Orkla Corn Plaster
Brief Title: A Clinical Investigation to Evaluate The Orkla Corn Plaster
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Orkla Care AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OCI-001
Record Dates: First submitted 2020-10-13; First posted 2020-10-23 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Corns
MeSH Terms: conditions — Callosities | interventions — Salicylic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Orkla corn plaster with Salicylic acid (Experimental)
  Interventions: Combination Product: Orkla Corn Plaster with salicylic acid
- Orkla corn protector without salicylic acid (Active Comparator)
  Interventions: Device: Orkla Corn Protector

INTERVENTIONS:
Combination Product: Orkla Corn Plaster with salicylic acid — Each participating subject will receive Orkla Corn Plasters for usage up to 28 days, or until corn resolution whichever comes first. Subjects will be instructed to change plasters daily.
  Arms: Orkla corn plaster with Salicylic acid
Device: Orkla Corn Protector — Each participating subject will receive Orkla Corn Protector for usage up to 28 days, or until corn resolution whichever comes first. Subjects will be instructed to change plasters daily.
  Arms: Orkla corn protector without salicylic acid

SUMMARY:
This is a prospective, randomized, controlled, open-labelled investigation to assess performance and safety of Orkla Corn Plaster in subject with corns. The hypothesis is that there is an improvement in the size of corns at day 28 compared to baseline.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form
2. >18 years of age
3. Presence of corn(s) confirmed by Investigator
4. Corn included into investigation shall not have been subject to any other treatment 1 month prior to study enrolment.

Exclusion Criteria:

1. Pregnant or lactating women at time of enrolment
2. Subjects with hypersensitivity to salicylic acid/salicylates, polyethylene foil, acrylic adhesive, viscose/polyethylene fibers and azorubine
3. Subjects diagnosed with diabetes
4. Subjects with poor peripheral blood circulation
5. Subjects with renal dysfunction (eGFR <60 mL/min/1.73 m2)
6. Subjects with ongoing skin disease in the area where the index corn is located.
7. Subjects with any other condition that as judged by the investigator may make follow-up or investigations procedures inappropriate
8. Any subject that according to the Declaration of Helsinki is unsuitable for enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2020-10-21 (Actual); Primary Completion 2021-01-14 (Actual); Study Completion 2021-06-10 (Actual)

PRIMARY OUTCOMES:
Percentage of improved subjects treated with Orkla Corn Plaster (with salicylic acid) at D28 compared to D0 (baseline) | 28 days

SECONDARY OUTCOMES:
Difference in percentage of improved subjects from D0 (baseline) to D28 between Orkla Corn Plaster (with salicylic acid) and Orkla Corn Protector (without salicylic acid) | 28 days
Percentage of improved subjects at D14, 3 and 6 months compared to baseline. | 14 days, 3 months and 6 months
  Comparisons within the Orkla Corn Plaster group, and comparison between the two treatment groups Orkla Corn Plaster vs. Orkla Corn Protector.
Pain experienced from index corn recorded on Visual Analog Scale (VAS; scale: 0-100 mm where a higher score corresponds to worse pain) at D14, D28, 3 and 6 months compared to baseline. | 14 days, 28 days, 3 months and 6 months
  Comparisons within the Orkla Corn Plaster group, and comparison between the two treatment groups Orkla Corn Plaster vs. Orkla Corn Protector.
Pain assessment recorded on Visual Analog Scale (VAS; scale: 0-100 mm where a higher score corresponds to worse pain) before and immediately after plaster application | Before and immediately after plaster application
  Comparisons within the Orkla Corn Plaster group, and comparison between the two treatment groups Orkla Corn Plaster vs. Orkla Corn Protector.
Resolution of corn at D14, D28, 3 and 6 months | 14 days, 28 days, 3 months and 6 months
  Comparisons within the Orkla Corn Plaster group, and comparison between the two treatment groups Orkla Corn Plaster vs. Orkla Corn Protector.
Subject reported resolution point of time (diary) | Up to 6 months
  Comparisons within the Orkla Corn Plaster group, and comparison between the two treatment groups Orkla Corn Plaster vs. Orkla Corn Protector.
Percentage of subjects with recurrence at D14, D28, 3 and 6 months | 14 days, 28 days, 3 months and 6 months
  Comparisons within the Orkla Corn Plaster group, and comparison between the two treatment groups Orkla Corn Plaster vs. Orkla Corn Protector.
Corn size reduction (mm) at D14, D28, 3 and 6 months | 14 days, 28 days, 3 months and 6 months
  Comparisons within the Orkla Corn Plaster group, and comparison between the two treatment groups Orkla Corn Plaster vs. Orkla Corn Protector.
Usability questionnaire: Ease of application assessed via subject-reported question with a 5-point qualitative scale. | 14 days, 28 days
  Percentage of subjects selecting a given answer is presented with comparisons within the Orkla Corn Plaster group, and comparisons between the two treatment groups, Orkla Corn Plaster vs. Orkla Corn Protector.
Usability questionnaire: Adherence to the application site assessed via subject-reported question with a 5-point qualitative scale. | 14 days, 28 days
  Percentage of subjects selecting a given answer is presented with comparisons within the Orkla Corn Plaster group, and comparisons between the two treatment groups, Orkla Corn Plaster vs. Orkla Corn Protector.
Subject treatment satisfaction questionnaire: Overall treatment satisfaction assessed via subject-reported question with a 5-point qualitative scale | 28 days
  Percentage of subjects selecting a given answer is presented with comparisons within the Orkla Corn Plaster group, and comparisons between the two treatment groups, Orkla Corn Plaster vs. Orkla Corn Protector.
Subject treatment satisfaction questionnaire: Corn appearance improvement assessed via subject-reported question with a 5-point qualitative scale | 28 days
  Percentage of subjects selecting a given answer is presented with comparisons within the Orkla Corn Plaster group, and comparisons between the two treatment groups, Orkla Corn Plaster vs. Orkla Corn Protector.
Subject treatment satisfaction questionnaire: Product recommendation assessed via subject-reported question with answer alternatives Yes/No/Don't know | 28 days
  Percentage of subjects selecting a given answer is presented with comparisons within the Orkla Corn Plaster group, and comparisons between the two treatment groups, Orkla Corn Plaster vs. Orkla Corn Protector.
Investigator treatment satisfaction questionnaire: Overall treatment satisfaction assessed via investigator-reported question with a 5-point qualitative scale | 28 days
  Percentage of subjects for each answer alternative (judged by investigator) is presented with comparisons within the Orkla Corn Plaster group, and comparisons between the two treatment groups, Orkla Corn Plaster vs. Orkla Corn Protector.
Investigator treatment satisfaction questionnaire: Corn appearance improvement assessed via investigator-reported questionnaire with a 5-point qualitative scale | 28 days
  Percentage of subjects for each answer alternative (judged by investigator) is presented with comparisons within the Orkla Corn Plaster group, and comparisons between the two treatment groups, Orkla Corn Plaster vs. Orkla Corn Protector.
Investigator treatment satisfaction questionnaire: Product recommendation assessed via investigator-reported questionnaire with answer alternatives Yes/No/Don't know | 28 days
  Percentage of subjects for each answer alternative (judged by investigator) is presented with comparisons within the Orkla Corn Plaster group, and comparisons between the two treatment groups, Orkla Corn Plaster vs. Orkla Corn Protector.

OTHER OUTCOMES:
Incidence of adverse events (AE), adverse device effects (ADE), serious adverse events (SAE), and serious adverse device effects (SADE), and device deficiency (DD) throughout the clinical investigation. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Felix Lundin, Principal Investigator — Carlanderska Hospital, Carlandersparken 1, 405 45 Göteborg, Sweden.
Locations (1):
- Carlanderska Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No